CLINICAL TRIAL: NCT00002196
Title: A Phase I Multiple Oral, Rising-Dose, Tolerance and Pharmacokinetic Trial of CI-1012 in HIV-1-Infected Volunteers.
Brief Title: A Study of CI-1012 in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parke-Davis (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 278A; 1012-005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Administration, Oral; Drug Administration Schedule; CD4 Lymphocyte Count; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: CI-1012

SUMMARY:
The purpose of this study is to see if it is safe and effective to give CI-1012 to HIV-infected patients who do not have any symptoms of the disease. This study also examines how the body handles CI-1012.

DETAILED DESCRIPTION:
Patients receive 2 weeks of oral CI-1012 therapy in this open-label study, with 8 patients entered at each dose level studied.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serologic evidence of infection with HIV-1.
* CD4+ cell count >= 200 cells/mm3.
* HIV-1 RNA >= 10,000 copies/ml.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

Viral, fungal, or bacterial infection requiring therapy other than topical medications.

Concurrent Medication:

Excluded:

* Prophylactic systematic antibacterial, antifungal or antiviral agents.
* Antiretroviral therapy. NOTE:
* Patient must be willing to remain off antiretroviral therapy for 1 week after completing study medication.

Prior Medication:

Excluded:

* Experimental therapy for >= 4 weeks prior to initiation of study medication.
* Antiretroviral treatment for 3 weeks prior to initiation of study medication.
* Systemic steroids or anticancer agents for 4 weeks prior to initiation of study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - ViRx Inc, Palm Springs, California
  - ViRx Inc, San Francisco, California
  - Central Florida Research Initiative, Maitland, Florida
  - Natl Institutes of Health, Bethesda, Maryland